CLINICAL TRIAL: NCT02857595
Title: Energy Balancing Modeling and Mobile Technology to Support e-Weight Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, John Graham Thomas, Associate Professor (Research), The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 212715 45CFR 46.110(4)(7)
Record Dates: First submitted 2016-08-02; First posted 2016-08-05 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (3):
- Online Weight Loss Program (Active Comparator)
  Interventions: Behavioral: Online Behavioral Weight Loss program
- Online Weight Loss Program + Nomogram (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss program; Behavioral: Weight Loss Nomogram
- Online Weight Loss Program + Nomogram + Bite Counter (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss program; Behavioral: Weight Loss Nomogram; Behavioral: Bite Counter

INTERVENTIONS:
Behavioral: Online Behavioral Weight Loss program
Behavioral: Weight Loss Nomogram
  Arms: Online Weight Loss Program + Nomogram; Online Weight Loss Program + Nomogram + Bite Counter
Behavioral: Bite Counter
  Arms: Online Weight Loss Program + Nomogram + Bite Counter

SUMMARY:
Behavioral lifestyle treatment for obesity produces clinically significant weight loss and corresponding improvements in disease risk and severity when delivered via in-person group and/or individual treatment sessions. Online versions have been developed in order to reduce costs. These programs typically include weekly weight loss lessons and tailored feedback on patients' weight loss progress. However, online programs often produce suboptimal outcomes compared to programs delivered in-person due to insufficient adherence to prescribed behavioral strategies, and a lack of objective methods for behavioral self-monitoring to support adherence. One approach to monitoring and improving adherence involves tracking patients' weight loss progress on a personalized nomogram (i.e., graph). The nomogram is based on a dynamic energy balance equation and depicts the expected weight loss over time if the participant is adherent to a prescribed goal for caloric intake and physical activity. A complementary approach to measuring and intervening on adherence involves the use of mobile technology to monitor eating behavior. The Bite Counter is a wrist-worn device similar to a wristwatch that measures the timing, frequency, rate, and duration of eating events by monitoring the "wrist roll" motion that occurs when food is brought to the mouth. By using mathematical models to "calibrate" the Bite Counter to the weight loss nomogram, it may be possible to identify the optimal number of bites that any given patient should take each day in order to facilitate weight loss. The purpose of the proposed study is to conduct a small randomized controlled trial to test the feasibility, acceptability, and preliminary efficacy of adding weight loss nomograms and the Bite Counter to an established online weight loss program. A sample of 30 participants with overweight/obesity will be randomly assigned in equal proportions to one of three 12-week weight loss programs: (a) online behavioral weight loss treatment alone (OBWL), (b) online behavioral weight loss treatment plus the provision of weight loss nomograms with weekly feedback tailored to the nomogram (OBWL+N), or (c) online behavioral weight loss treatment plus the provision of weight loss nomograms with weekly feedback tailored to the nomogram and provision of a Bite Counter that can be used to alert participants when they are approaching their maximum number of prescribed bites per day (OBWL+N&BC).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 27 and 45 kg/m^2

Exclusion Criteria:

* Self-report of health problems that make weight loss or unsupervised exercise unsafe or unreasonable
* A heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire
* Currently pregnant or intend to become pregnant in the next 6 months
* Planning to move outside of the geographic region within the next 6 months
* Self-report any cognitive or physical limitations that preclude use of a personal computer
* Participation in a study conducted at the research center in the past 2 years
* Use of a commercial weight loss program within the last 6 months
* Self-report a history of clinically diagnosed eating disorder excluding Binge Eating Disorder
* Previous surgical procedure for weight loss
* Current use of weight loss medication
* Treatment of cancer within the last 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Weight Loss | 6 months after beginning treatment

SECONDARY OUTCOMES:
Number of online weight loss lessons viewed | 6 months after beginning treatment
Number of weeks body weight, caloric intake, and physical activity reported online | 6 months after beginning treatment
Number of weekly clinic visits attended | 6 months after beginning treatment
Average number of bites of food per day | 6 months after beginning treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Miriam Hospital Weight Control and Diabetes Resarch Center, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Goldstein CM, Goldstein SP, Thomas DM, Hoover A, Bond DS, Thomas JG. The Behavioral Intervention with Technology for E-Weight Loss Study (BITES): Incorporating Energy Balance Models and the Bite Counter into an Online Behavioral Weight Loss Program. J Technol Behav Sci. 2021 Jun;6(2):406-418. doi: 10.1007/s41347-020-00181-4. Epub 2020 Nov 27. PMID 35356149